CLINICAL TRIAL: NCT02846571
Title: Pancreatic Islet Transplantation Into the Anterior Chamber of the Eye
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Midhat H. Abdulreda (Other)
Collaborators: Diabetes Research Institute Foundation (Other); Bascom Palmer Eye Institute (Other)
Responsible Party: Sponsor-Investigator, Midhat H. Abdulreda, Associate Professor, Diabetes Research Institute, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160640
Record Dates: First submitted 2016-07-18; First posted 2016-07-27 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Diabetes
Keywords: Islet Transplantation; Type 1 Diabetes; Immune Tolerance Induction; Diabetes Complications; Intraocular Transplantation; Eye Anterior Chamber; Kidney Transplantation; Immunosuppression; Type 2 Diabetes; Eye Drops Immunosuppression; localized immunosuppression
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Complications; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Human Pancreatic Islet Transplantation (Other): Islet transplantation into the anterior chamber of the eye single arm
  Interventions: Biological: Human Pancreatic Islet Transplantation

INTERVENTIONS:
Biological: Human Pancreatic Islet Transplantation — Human pancreatic islet transplantation in the eye anterior chamber of legally blind type 1 or type 2 diabetes patients with and without insulin-dependence

SUMMARY:
The intervention in this trial is intraocular islet transplantation. A single dose of 1000 - 3000 Islet Equivalents (IEQ)/kg recipient body weight (BW) will be infused into the anterior chamber of the eye through a self-sealing incision in the peripheral cornea. The procedure is projected to take approximately 20-30 minutes. Subject will remain flat on their back for 1 - 3 hours after islet infusion to maximize adhesion of the islets to the iris.

DETAILED DESCRIPTION:
The American Diabetes Association reports that 38.4 million Americans had diabetes in 2021, which accounts for 11.6% of the population. About 77% of them were diagnosed (29.7 million) and the rest were undiagnosed (8.7 million). With an estimated 1.2 million new diagnoses every year, the number of people living with diabetes in the U.S. alone is estimated to increase by the end of the decade to 45.6 million. Approximately 95% of diabetics have type 2 diabetes (T2D) and the rest (~2 million) are type 1 diabetics (T1D); although, the prevalence of T1D is also increasing. According to the Juvenile Diabetes research Foundation (JDFR), an anticipated 64,000 new T1D diagnoses are expected each year in the U.S., and similar trends have been observed in children and adolescents in many other countries. Consequently, the combined global economic cost of diabetes healthcare is expected to be around $2.2 trillion by 2030.

While the etiologies of T1D and T2D may vary, both can lead to insulin insufficiency and hyperglycemia (increased blood sugar levels). Chronic hyperglycemia results in diabetic complications that severely impact on the quality-of-life of patients and some can be life-threatening, like diabetic ketoacidosis. Therefore, insulin supplementation in insulin-dependent diabetes is required. Insulin supplementation can be either in the form of multiple daily insulin injections (manual or via pump) or by biological replacement of the insulin-producing beta cells through transplantation, which provides a natural source of insulin. On the one hand, since the discovery of insulin in the early 1900s, exogenous insulin supplementation has saved countless lives of diabetic patients. However, it is well established that exogenous insulin injection therapy is suboptimal in preventing fluctuation in blood sugar levels (i.e., hyper- and hypoglycemia) due to mis-dosing and other factors. On the other hand, transplantation provides an endogenous source of insulin and c-peptide in real-time without the need for pre-meal dosing or the risk of miscalculating the dose in manual administration or for the challenging predictive algorithms in the case of insulin pumps. Importantly, it has been shown that even partial levels of endogenous insulin secretion can improve glycemic lability and protect from chronic diabetic complications and life-threatening hypoglycemia and diabetic ketoacidosis.

It is now established that beta cell replacement therapy through transplantation of isolated pancreatic islets offers a great therapeutic option in insulin-dependent diabetes, and FDA recently approved it as the first cellular therapy in T1D. However, islet transplantation also has limitations. In general, the limited availability of donor tissue remains a significant obstacle in transplant therapies, including that of pancreatic islets. Other limitations are associated with the mandatory use of systemic anti-rejection immunosuppressive drugs because chronic systemic immunosuppression exposes the transplant recipients to serious and potentially deadly side-effects and complications, such as, but not limited to, increased susceptibility to infections, sepsis, and cancer. While improving systemic immunosuppression regimens would reduce off-target effects and the associated systemic complications, avoiding generalized immunosuppression altogether via localized application would significantly reduce such undesired complications.

Currently, diabetic patients receive transplant therapy either in the form of whole pancreas or isolated pancreatic islets. On the one hand, whole pancreas transplant has been shown to achieve insulin independence in T1D patients, but it is also very invasive and is associated with a high risk of complications and adverse events including mortality. On the other hand, transplantation of isolated pancreatic islets is minimally invasive and has significantly less complications compared to whole pancreas transplant, but survival of the islet graft might be severely limited by complications associated with the current clinical transplant site, the portal system of the liver. Nevertheless, thousands of patients have received islet transplants in their livers in clinical trials that demonstrated its benefits and the significant improvement in the quality-of-life of islet transplant recipients brought about through improved glycemic control, reduced hypoglycemia episodes, and the prevention of diabetes-associated complications. Notably, some transplanted patients with restored awareness of hypoglycemia maintained this benefit even after going back on exogenous insulin therapy due to islet-graft loss. Many transplant recipients with diabetic retinopathy (D.R.) also experienced improvement in their D.R. Recent experimental evidence indicates that this improvement is mediated by c-peptide inhibiting VEGF-induced vasculopathies, which occur in both T1D and T2D patients. Therefore, transplantation of pancreatic islets is a good treatment option in insulin-dependent diabetes.

The current trial is evaluating the safety of intraocular islet transplantation with localized maintenance immunosuppression via topical application of eye-drops.

ELIGIBILITY:
Patients who meet all of the following criteria are eligible for participation in the study:

Ophthalmic inclusion criteria:

1. Patient with at least one eye with extensive loss of vision from hand motion to no light perception.
2. Phakic or pseudophakic with a stable intraocular lens in the blind eye.
3. Normal cornea with good visualization of the anterior segment.
4. Normal anterior segment anatomy including the iris bed.

General and metabolic inclusion criteria:

1. Male and female subjects ages 18 to 75 years of age and no history of non-compliance.
2. Clinical history compatible with T1D or T2D with or without insulin-dependence at the time of enrollment.
3. Stable renal function of native or transplanted kidney if applicable.
4. Ability to provide written informed consent.
5. Mentally stable and able to comply with the procedures of the study protocol.

Exclusion Criteria: Patients who meet any of these criteria are not eligible for participation in the study:

Ophthalmic exclusion criteria (only in surgical eye):

1. Poor visualization of the anterior chamber (corneal opacity, corneal edema, Herpes Keratitis).
2. Aphakic status (no lens).
3. Narrow angle of iris anatomy: Spade Scale IV.
4. History of uncontrolled glaucoma or glaucoma that had required surgical intervention (e.g., trabeculectomy or shunting devices).
5. Active uncontrolled uveitis.
6. Presence of silicone in the anterior segment after complex diabetic retinopathy surgery.
7. History of allergy to topical steroids and immune-modulatory drugs including CSA and Tacrolimus.

General and metabolic exclusion criteria:

1. HbA1c >10%.
2. Blood Pressure: SBP >160 mmHg or DBP >100 mmHg.
3. Calculated GFR of ≤40 mL/min/1.73 m2 for patients with kidney transplant or <80 mL/min/1.73 m2 for those without kidney transplant, using the subject's measured serum creatinine and the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation1.
4. Strict vegetarians (vegans) will be excluded only if their estimated GFR is ≤35 mL/min/1.73 m2 for patients with kidney transplant or <70 mL/min/1.73 m2 for those without kidney transplant.
5. Proteinuria (albumin/creatinine ratio or ACr >300mg/dl) of new onset or since kidney transplantation if applicable.
6. Calculated panel-reactive anti-HLA antibodies >20%.
7. Positive crossmatch.
8. Antibodies (i.e., presumed de-novo) to the kidney transplant donor, if applicable.
9. For female subjects: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study (24 months) or within 4 months after discontinuation, or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
10. Presence or history of active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB). Subjects with laboratory evidence of active infection are excluded even in the absence of clinical evidence of active infection.
11. Negative screen for Epstein-Barr Virus (EBV) by IgG determination.
12. Invasive aspergillus, histoplasmosis, and coccidioidomycosis infection within one year prior to study enrollment.
13. Active malignancy (cancer) except if successfully treated and declared cancer-free and/or in-remission by the oncologist.
14. Known active alcohol or substance abuse.
15. Baseline Hb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/µL), neutropenia (<1,500/µL), or thrombocytopenia (platelets <100,000/µL). Participants with lymphopenia are allowed if the investigator determines there is no additional risk with additional clearance from a hematologist.
16. Severe co-existing cardiac disease, characterized by any one of these conditions:

    1. Recent myocardial infarction (within past 6 months).
    2. Evidence of ischemia on functional cardiac exam within the last year.
    3. Left ventricular ejection fraction <30%.
17. Hyperlipidemia despite medical therapy (fasting low-density lipoprotein [LDL] cholesterol >130 mg/dL, treated or untreated; and/or fasting triglycerides >200 mg/dL).
18. Receiving treatment for a medical condition requiring chronic use of systemic steroids, except for the use of ≤5 mg prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only.
19. Use of any investigational agents within 4 weeks of enrollment.
20. Administration of live attenuated vaccine(s) within 2 months of enrollment.
21. Any medical condition that, in the opinion of the investigator, will interfere with the safe participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Absence of ocular complications | 24 months after transplant
  Absence of, corneal decompensation, increased intraocular pressure (IOP), uveitis, cataract formation, retinal detachment, retinal bleeding, retinal vasculopathies, macular edema, optic neuropathy, and endophthalmitis in the transplanted eye
Absence of sympathetic ophthalmia | 24 months after transplant
  Absence of ophthalmic complications in the non-transplanted eye and assessment of diabetic retinopathy compared to baseline before transplant
Confirmation of intraocular islet graft survival | 24 months after transplant
  Confirmation of positive c-peptide (>1 ng/ml) in the aqueous humor of the transplanted eye and assessment of intraocular islet graft integrity by slit-lamp microscopy and OCT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Midhat H Abdulreda, Ph.D., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Bascom Palmer Eye Institute, Miami, Florida
  - Diabetes Research Institute, University of Miami Miller School of Medicine, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez VL, Caicedo A, Berman DM, Arrieta E, Abdulreda MH, Rodriguez-Diaz R, Pileggi A, Hernandez E, Dubovy SR, Parel JM, Ricordi C, Kenyon NM, Kenyon NS, Berggren PO. The anterior chamber of the eye as a clinical transplantation site for the treatment of diabetes: a study in a baboon model of diabetes. Diabetologia. 2011 May;54(5):1121-6. doi: 10.1007/s00125-011-2091-y. Epub 2011 Mar 1. PMID 21360190
- [Background] Shishido A, Caicedo A, Rodriguez-Diaz R, Pileggi A, Berggren PO, Abdulreda MH. Clinical intraocular islet transplantation is not a number issue. CellR4 Repair Replace Regen Reprogram. 2016;4(4):e2120. Epub 2016 Jul 26. PMID 29497631
- [Background] Tun SBB, Chua M, Hasan R, Kohler M, Zheng X, Ali Y, Abdulreda MH, Juntti-Berggren L, Barathi VA, Berggren PO. Islet Transplantation to the Anterior Chamber of the Eye-A Future Treatment Option for Insulin-Deficient Type-2 Diabetics? A Case Report from a Nonhuman Type-2 Diabetic Primate. Cell Transplant. 2020 Jan-Dec;29:963689720913256. doi: 10.1177/0963689720913256. PMID 32264703
- [Background] Abdulreda MH, Berman DM, Shishido A, Martin C, Hossameldin M, Tschiggfrie A, Hernandez LF, Hernandez A, Ricordi C, Parel JM, Jankowska-Gan E, Burlingham WJ, Arrieta-Quintero EA, Perez VL, Kenyon NS, Berggren PO. Operational immune tolerance towards transplanted allogeneic pancreatic islets in mice and a non-human primate. Diabetologia. 2019 May;62(5):811-821. doi: 10.1007/s00125-019-4814-4. Epub 2019 Jan 31. PMID 30701283
- See also: CellR4 Publication — http://www.cellr4.org/article/2120